# CLINICAL STUDY PROTOCOL AMENDMENT

# A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Phase 2a Study to Determine Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Activity of NFX-179 Gel in Subjects with Cutaneous Neurofibromas

| Protocol No. | NFX-179-NF1-201 |
|---|---|
| Protocol/Amendment Date: | 01-APR-2021 |
| Amendment No.: | 3 |
| Supersedes: | N/A |
| Sponsor: | NFlection Therapeutics 714 Woodcrest Road, Wayne, PA 19087 United States |
| | Guy Webster, M.D. Ph.D. 24-hour telephone: (302) 559-8684 Email: GWebster@Nflectionrx.com |

#### CONFIDENTIALITY STATEMENT

This document contains proprietary and confidential information of NFlection Therapeutics. Acceptance of this document constitutes agreement by the recipient that no previously unpublished information contained herein will be published or disclosed without the prior written approval of NFlection Therapeutics with the exception that this document may be disclosed to study staff under your supervision who need to know the contents for conducting the study and to appropriate Institutional Review Boards /Ethics Committees under the condition that the staff have agreed to keep this information confidential. The foregoing shall not apply to disclosure required by governmental regulations or laws, however, NFlection Therapeutics shall be promptly notified of any such disclosure.

Date: 01-APR-2021 Page 1 of 5 Supersedes: NEW

# PROTOCOL AMENDMENT INVESTIGATOR SIGNATURE PAGE

Protocol Number: NFX-179-NF1-201 Amendment Number: 3

#### **INVESTIGATOR COMMITMENT:**

I will provide copies of the protocol, any subsequent protocol amendments and access to all information provided by NFlection to the investigational center staff under my supervision. I will discuss this material with them to ensure that they are fully informed about the Investigational Medicinal Product and the study protocol.

I agree to conduct this clinical study according to the attached protocol, except when mutually agreed to with NFlection in writing. I also agree to conduct this study in compliance with all local regulatory requirements, Good Clinical Practices, as well as with the requirements of the appropriate Institutional Review Board(s) /Ethics Committee(s) and any other Institutional requirements.

| rinted Name of Investigator |
|-----------------------------|
| gnature of Investigator |
| ate |

Date: 01-APR-2021 Page 2 of 5 Supersedes: NEW

# PROTOCOL AMENDMENT APPROVAL PAGE

Protocol Number: NFX-179-NF1-201 Amendment Number: 3

A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Phase 2a Study to Determine Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Activity of NFX-179 Gel in Subjects with Cutaneous Neurofibromas

| Protocol No. | NFX-179-NF1-201 |
|---|---|
| Protocol/Amendment Date: | 01-APR-2021 |
| Amendment No.: | 3 |
| Sponsor: | NFlection Therapeutics<br>714 Woodcrest Road,<br>Wayne, PA 19087<br>United States |

C. Colo

04-02-2021

Christopher Powala Chief Executive Officer NFlection Therapeutics

Date

Guy Webster, M.D., Ph.D. Chief Medical Officer NFlection Therapeutics

Date

# **TABLE OF CONTENTS**

| <b>PROT</b> | OCOL AMENDMENT INVESTIGATOR SIGNATURE PAGE | 2 |
|-------------|--------------------------------------------|----|
| PROT | OCOL Amendment APPROVAL PAGE | 3 |
| | E OF CONTENTS | |
| | AMENDMENT HISTORY | |
| | AMENDMENT SUMMARY | |
| | AMENDMENT RATIONALE | |
| | PROTOCOL CHANGES. | |
| 4 | TRUTUCUL CHANGES | -2 |

#### 1 AMENDMENT HISTORY

Revised protocol 1 footer date: 24-JUL-2020

Previous amendments: Amendment 2, footer date 25-MAR-2021

#### 2 AMENDMENT SUMMARY

The following section of the NFX-179-NF1-201 revised protocol (footer date 24-JUL-2020) as modified by amendment 2 (footer date 25-MAR-2021) and with a final NFlection Therapeutics approval signature date of 27-JUL-2020 is amended:

• Section 8.3.3 Efficacy analyses.

# 3 AMENDMENT RATIONALE

This protocol change is made to allow for Target cNF Tumors that are found not to be qualifying neurofibromas to be excluded from sensitivity analyses of efficacy results.

# 4 PROTOCOL CHANGES

# Section 8.3.3 Efficacy analyses:

# Previous paragraph 1:

"...Tumor volume is the primary measurement of interest; however, the ruler measurements of tumor length and height will also be analyzed as described below."

# Changed paragraph 1:

"...Tumor volume is the primary measurement of interest; however, the ruler measurements of tumor length and height will also be analyzed as described below. Any Target cNF Tumors confirmed not to be qualifying neurofibromas based on histological evaluation of the excised tissue may be excluded from sensitivity analyses of efficacy results."